CLINICAL TRIAL: NCT03478761
Title: 24-Hydroxylase Deficiency and CYP24A1 Mutation Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David J. Sas, Principal Investigator, Mayo Clinic
Other Study IDs: 17-003972
Record Dates: First submitted 2018-03-22; First posted 2018-03-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: 24-hydroxylase Deficiency
Keywords: CYP24A1 mutation; CYP24A1; 24-hydroxylase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 24,25 Vitamin D testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
You are being asked to take part in this research registry because you or your family member is suspected to have a 24-hydroxylase deficiency.

DETAILED DESCRIPTION:
In this registry we propose to establish and maintain a registry of suspected and confirmed patients with 24 hydroxylase deficiency in an effort to collect data for further investigation. This would be the first and only known registry of its kind. These resources would be made widely available to clinicians and research scientists within Mayo to stimulate advances in the diagnosis and treatment of patients with this disease.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone genetic testing for a CYP24A1 mutation with at least 3 of the following:

* Urinary Stone Disease
* Nephrocalcinosis
* Metabolic Bone Disease
* Serum Calcium >/= 9.6 mg/dL
* Parathyroid hormone (PTH) < 30 pg/mL
* 1,25-dihydroxyvitamin D > 40 pg/mL OR a family member of a patient who meets the above criteria

Exclusion Criteria:

Patients who have tested negative for a CYP24A1 mutation with an alternative diagnosis that might explain hypercalcemia/hypercalciuria/stone disease:

* Sarcoidosis
* Lymphoma
* Tuberculosis
* Fungal infections
* Excessive exogenous calcium or vitamin D intake

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 24-hydroxylase deficiency and CYP24A1 mutation patient
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
establish and maintain a registry of suspected and confirmed patients with 24 hydroxylase deficiency | yearly
  This patient registry will expand knowledge of the clinical expression of this disease by systematically accumulating and analyzing information regarding a larger number of patients than have been studied to date.

SECONDARY OUTCOMES:
Improved understanding of symptoms and progression of this disease | yearly
  The goal of the patient registry is to collect data about this rare diseases, provide a better understanding of this conditions and help to develop new treatments.

CONTACTS AND LOCATIONS:
Overall Officials: David Sas, MD, Principal Investigator — Mayo Clinic; Peter Tebben, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials